CLINICAL TRIAL: NCT07095842
Title: Efficacy of Add-on Ketamine With Second-dose Midazolam for Prehospital Treatment of Epileptic Children With Status Epilepticus
Brief Title: Prehospital Early Administration of Ketamine for Status Epilepticus in Epileptic Kids (PEAK-SEEK)
Acronym: PEAK-SEEK
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Elsayed Abdelkreem, Assistant Professor of Pediatrics, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-25-7-4PD
Record Dates: First submitted 2025-07-23; First posted 2025-07-31 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Convulsive Status EPILEPTICUS
MeSH Terms: conditions — Status Epilepticus | interventions — Ketamine; Midazolam

STUDY DESIGN:
Intervention Model Description: This is a pragmatic, decentralized, pre-consented, event-driven randomized controlled trial. The investigators aim to recruit and pre-randomize up to 668 patients who meet the eligibility criteria. These participants will be randomized to receive either add-on intramuscular ketamine combined with a second dose of midazolam, or a second dose of midazolam alone, in the event of convulsive status epilepticus (CSE) that is not terminated by an initial dose of midazolam. The sample size has been calculated to ensure that approximately 100 participants will experience the qualifying event (CSE not responding to first-dose midazolam) and receive the assigned study medications, anticipating that 50 will receive ketamine plus second-dose midazolam and 50 will receive the second dose of midazolam alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine + Midazolam (Experimental)
  Interventions: Drug: Ketamine; Drug: Midazolam
- Midazolam (Active Comparator)
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — Intramuscular ketamine 2 mg/kg (max 90 mg)
  Arms: Ketamine + Midazolam
Drug: Midazolam — Intramuscular midazolam 0.2 mg/kg (max 10 mg)

SUMMARY:
The goal of this pragmatic, decentralized, pre-consented, event-driven, randomized controlled trial is to investigate the efficacy of add-on ketamine to second-dose midazolam for prehospital treatment of epileptic children with convulsive status epilepticus.

DETAILED DESCRIPTION:
Status epilepticus (SE) is the most prevalent neurological emergency in children. Benzodiazepines (BDZs) remain the first-line anti-seizure medication (ASM) for SE, but about one-third of seizures are not controlled by BDZs. Moreover, second-line ASMs (levetiracetam, valproate, phenytoin) fail to terminate BDZ-refractory SE in 50% of cases. Such prolonged SE is linked with progressive brain damage and an increased risk of epilepsy, irreversible neurodevelopmental sequelae, and mortality. Accordingly, early control of SE is critical for enhancing clinical outcomes.

A possible strategy for rapid control of SE is using early ASM combination. Ketamine seems a promising choice for such a combination. Ketamine acts to antagonize N-methyl-D-aspartate (NMDA) receptors, which become increasingly upregulated and trafficked to the synaptic membrane during ongoing seizure activity. Numerous observational studies have demonstrated that administration of ketamine is associated with termination or attenuation of refractory SE (RSE) and super-refractory SE (SRSE). Furthermore, the recently published Ket-Mid study showed that the ketamine-midazolam combination was more effective than midazolam alone in the initial treatment of pediatric generalized CSE. However, the Ket-Mid study also highlighted a significant delay in hospital arrival and administration of first-line ASM, by a median of 34 minutes, reflecting delayed access to emergency care due to socioeconomic challenges, geographic barriers, and limited prehospital emergency medical services. Such a challenge also applies to resource-limited settings, where treatment delays are more common. Notably, a review by Gaínza-Lein et al. of 15 studies involving 2212 patients with SE reported average times to ASM treatment and hospital arrival of 42.4 and 56 minutes, respectively. Such delay to the administration of ASM is associated with increased resistance to BZDs, longer SE, and increased risk of complications. Accordingly, there is a growing interest in the early use of ASM for prehospital treatment of SE.

Ketamine has been used in prehospital setting for a long time, mainly for sedation and analgesia purposes with a high safety profile. Multiple observational studies have reported the efficacy of ketamine in the pre-hospital emergency treatment of BZD-refractory status epilepticus. However, this was not adequately investigated in clinical trials.

The present study (Prehospital Early Administration of Ketamine for Status Epilepticus in Epileptic Kids, PEAK-SEEK) aims to investigate the efficacy of adding ketamine to second-dose midazolam vs. second-dose midazolam alone as ASM for prehospital treatment of epileptic children with convulsive status epilepticus.

ELIGIBILITY:
Inclusion Criteria:

* Age from 2 to 16 years.
* Established diagnosis of epilepsy of at least 1 year duration.
* History of at least 1 episode of convulsive status epilepticus in the preceding 12 months.

Exclusion Criteria:

* Failure to obtain informed consent.
* Known allergies or contraindications to ketamine.
* Known contraindications to intramuscular injection.
* Presence of another family member included in the same trial.
* Having subsequent events (only the index event will be included).

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 668 (Estimated)
Dates: Start 2025-08-03 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with cessation of seizures at the time of hospital arrival | At the time of hospital arrival (up to 1 hour)
  Number of participants with cessation of clinically evident seizures at the time of hospital arrival

SECONDARY OUTCOMES:
Number of participants with sustained cessation of seizures | From 10 minutes after study drug administration to 60-minutes after hospital arrival
  Number of participants with sustained cessation of clinically evident seizures at 10 minutes after study drug administration to 60-min after hospital arrival with improved responsiveness (verbal communication, obeying commands, or purposeful reaction to painful stimuli) and no endotracheal intubation or use of any additional antiseizure medications or anticonvulsant sedatives
Number of participants with recurrence of seizures | From 10 minutes after study drug administration to 60-minutes after hospital arrival
  Number of participants with recurrence of clinically evident seizures after initial control at 10 minutes after study drug adminstration till 60-minutes after hospital arrival
Number of participants underwent endotracheal intubation | 60 minutes after hospital arrival
  Number of participants underwent endotracheal intubation at 60 minutes after hospital arrival
Number of participants with severe hypotension | At the time of hospital arrival (up to 1 hour)
  Number of participants with severe hypotension at the time of hospital arrival
Number of participants with severe hypertension | At the time of hospital arrival (up to 1 hour)
  Number of participants with severe hypertension at the time of hospital arrival
Number of participants with severe cardiac arrhythmia | At the time of hospital arrival (up to 1 hour)
  Number of participants with severe cardiac arrhythmia at the time of hospital arrival
Number of participants with emergence reactions | At the time of hospital arrival (up to 1 hour)
  Number of participants with emergence reactions (hallucination, delirium, vivid dreams, blurred/double vision, hypersalivation) following study drug administration till hospital arrival

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics at Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No
Unidentified individual participant data will be available to qualifying researchers upon a reasonable request